CLINICAL TRIAL: NCT06928623
Title: Anxiety in Non-professional Football Players With Recurrent Hamstring Injuries. An Ambispective Cohort Study.
Brief Title: Anxiety in Non-professional Football Players With Recurrent Hamstring Injuries.
Status: Not yet recruiting | Type: Observational
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Rubén Cuesta-Barriuso, PhD, Principal Investigator, Universidad Católica San Antonio de Murcia
Other Study IDs: AnsFut
Record Dates: First submitted 2025-03-31; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Football Player
Keywords: Football players; Anxiety; Hamstring muscles; Recurrence of injury; Physiotherapy
MeSH Terms: conditions — Anxiety Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group: A single measurement will be taken, and the data will be analyzed anonymously, as the identity of the patients filling in the questionnaires will be unknown to the analyst. The primary variable of the study will be anxiety, with the number of recurrences of the lesion under study being the dependent variable. The secondary variables, estimated as modifying or confounding variables, will be the main clinical, sports, anthropometric and sociodemographic variables.
  Interventions: Other: Surveys

INTERVENTIONS:
Other: Surveys — In the present study, no intervention will be carried out, with the recruited subjects only completing the questionnaires set out in the study variables.

SUMMARY:
Introduction. Faced with the risk of injury relapse, and as athletes train and compete, they generate anxiety that limits their ability to push themselves to the maximum, influencing their performance.

Objectives. i) To identify the state and trait anxiety of non-professional athletes with previous hamstring injuries; ii) To evaluate the main prognostic factors of anxiety in these athletes; and iii) To analyze the best predictive model of anxiety in soccer players with previous hamstring injuries.

Material and method. Ambispective cross-sectional cohort study. 88 players will be recruited. The primary variable of the study will be anxiety (State-Trait Anxiety Inventory), with the number of recurrences of the study injury being the dependent variable. The secondary variables, estimated as modifying or confounding, will be the main sociodemographic variables (age, type of school/work activity), clinical (number of hamstring injuries, number of relapses of injury in the same location, duration of injury in weeks, date of last injury), sports (weekly training load, seasons competing, regular starting line-up) and anthropometric (weight).

ELIGIBILITY:
Inclusion Criteria:

* Male athletes aged 18 to 19
* Registered in the Division of Honor category of the Region of Murcia
* Who are university students
* With previous hamstring injuries in the last 12 months.

Exclusion Criteria:

* Athletes with an injury, muscular or not, at the time of the study
* Athletes in their first year as registered soccer players.

Ages: 18 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Footballers who will be recruited to the teams Real Murcia, Real Murcia Promesas, Alcantarilla, UCAM, Churra, Guadalupe, all of them belonging to the under-19 category.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2025-04-29 (Estimated); Study Completion 2025-05-25 (Estimated)

PRIMARY OUTCOMES:
Assessment of anxiety | Screening visit
  Anxiety will be evaluated using the State-Trait Anxiety Inventory. This scale will be used to measure the perception of anxiety of the patients included in the study. The state and trait of anxiety of each subject is evaluated with a score of 0 to 30 points for each scale, where a higher score indicates a higher anxiety index in the trait or state.

SECONDARY OUTCOMES:
Assessment of the main sociodemographic variables | Screening visit
  In the evaluation of the main sociodemographic variables, the following will be evaluated: age (in completed months) and type of school/work activity (sedentary/active)
Measuring the number of hamstring injuries | Screening visit
  For the data analysis, each subject will be asked to indicate, among the clinical variables, the number of hamstring injuries they have had over the last 3 seasons
Measurement of weekly training load | Screening visit
  For the data analysis, each subject will be asked to indicate, among the sports variables, the weekly training load (in hours) that they usually have during the competition stage of the season.
Assessment of the main anthropometric variables | Screening visit
  In the assessment of the main anthropometric variables, weight (in kg) will be measured.
Measuring the duration of hamstring injuries | Screening visit
  For the data analysis, each subject will be asked to indicate, among the clinical variables, the duration (measured in weeks) of the hamstring injuries they have had over the last 3 seasons
Measurement of the date of the last hamstring injury | Screening visit
  For the data analysis, each subject will be asked to indicate, among the clinical variables, the date of the last injury (measured in weeks) to the hamstring muscles over the last 3 seasons
Measurement of the number of seasons that the soccer player has been competing | Screening visit
  For the data analysis, each subject will be asked to indicate, among the sports variables, the number of seasons that they have been federated, competing in soccer.
Measurement of the footballer's regular starting position in the team | Screening visit
  For the data analysis, each subject will be asked to indicate, among the sporting variables, the footballer's regular starting position in the football team, with a dichotomous answer (yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, Principal Investigator — Universidad de Oviedo

IPD SHARING:
Plan to Share IPD: Undecided